CLINICAL TRIAL: NCT06866925
Title: Transcranial Direct Current Stimulation as a Treatment for Depression With Catatonic Features in Patients With Down Syndrome: a Pilot Randomized Sham-controlled Study
Brief Title: tDCS for Catatonic Depression in Down Syndrome: A Pilot Study
Acronym: TOTORO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-A00452-45; PHRC-23-0027 (Other Grant/Funding Number: DGOS)
Record Dates: First submitted 2025-02-26; First posted 2025-03-10 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Down Syndrome
Keywords: catatonia
MeSH Terms: conditions — Down Syndrome; Catatonia

STUDY DESIGN:
Intervention Model Description: Multicenter (6 sites), randomized, double-blind, parallel-group controlled study. Patients will be randomly assigned to a group receiving 15 sessions of active tDCS (3 sessions per day for 5 days, from D0 to D5, with the tDCS anode placed over the left DLPFC and the cathode over the right DLPFC, located using the international 10/20 electrode placement system, each stimulation lasting 20 minutes at 2mA), or to a group receiving 15 sessions of sham stimulation (same electrode montage and stimulation duration, but without current). Participation in the EEG and biology component will be limited to the Lyon and Paris centers.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS (Active Comparator): Group receiving 15 sessions of active tDCS (3 sessions per day for 5 days, from D0 to D5, with the tDCS anode placed over the left DLPFC and the cathode over the right DLPFC, located using the international 10/20 electrode placement system, each stimulation lasting 20 minutes at 2mA).
  Interventions: Device: Transcranial stimulation
- Sham tDCS (Placebo Comparator): Group receiving 15 sessions of sham stimulation (same electrode montage and stimulation duration, but without current).
  Interventions: Device: Transcranial stimulation

INTERVENTIONS:
Device: Transcranial stimulation — A randomized, 2-arm, sham-controlled study, patients with Down syndrome presenting with major depressive episode (DSM5) with catatonic features will be randomly allocated to receive 15 sessions of either active (20 min, 2mA, ramp up/down 30 sec) or sham tDCS (20 min, ramp up/down 30 sec at the beginning and at the end of each stimulation session), thrice daily. Each stimulation session will be spaced at least two hours apart. The anode will be placed over the left DLPFC, the cathode over the right DLPFC using the Beam F3 algorithm in order to individualize target location based on head circumference, tragus to tragus and inion to nasion distances.

SUMMARY:
This study evaluates the efficacy of transcranial direct current stimulation (tDCS) for depression with catatonia in individuals with Down syndrome (DS). 62 patients will be randomized to receive 15 sessions of active or sham tDCS. The primary objective is to measure changes in depressive/catatonic symptoms using the Bush-Francis Catatonia Rating Scale (BFCRS). Secondary objectives include safety, cognitive effects, EEG correlates, and biological markers (cortisol, BDNF, cytokines). The study aims to provide a non-pharmacological therapeutic alternative for this population

DETAILED DESCRIPTION:
Justification: Depression is common in individuals with Down syndrome (DS), often accompanied by catatonia, and is under-treated. Conventional treatments are limited by tolerability and linguistic difficulties. Transcranial direct current stimulation (tDCS), safe and effective, has never been tested in DS.

Hypothesis: tDCS is effective and safe for depression with catatonia in DS, improving mood, cognition, and motor symptoms.

Objectives:

Primary: To evaluate the clinical efficacy of 15 sessions of bifrontal tDCS on depression with catatonia in DS (Bush-Francis Catatonia Rating Scale (BFCRS)).

Secondary: To evaluate safety, long-term clinical and cognitive effects (1 and 3 months), EEG correlates, and biological effects (cortisol, BDNF, cytokines).

Methodology: Multicenter (2 sites), randomized, double-blind, placebo-controlled study. 30 DS patients will receive 15 sessions of active tDCS (2 mA, 20 min, anode over left DLPFC, cathode over right DLPFC) or sham tDCS.

Outcomes:

Primary: Changes in depressive/catatonic symptoms (BFCRS) between Day 0 and Day 5.

Secondary: Safety, clinical (MADRS, UPDRS), cognitive (SIB), EEG, and biological (blood, saliva) assessments.

Target Population: Men and women with DS with a depressive episode and catatonia (30 patients).

Inclusion Criteria: DS, age > 18 years, major depression with catatonia (DSM-5), informed consent.

Exclusion Criteria: Pregnancy, contraindication to tDCS, refusal. Statistical Analyses: ANOVA or mixed models for BFCRS scores. Justification for Inclusion: To provide a safe, non-pharmacological therapeutic alternative.

Withdrawal Criteria: Withdrawal of consent, severe pathology. Procedures: Clinical, cognitive, EEG, and biological (blood, saliva) assessments at Day 0, Day 1, Day 5, 1 and 3 months.

Recruitment: 6 sites (CH Vinatier Lyon, CHU Nantes, CHU Dijon, CHU Clermont Ferrand, CH Rouen, GHU Neurosciences Paris). EEG and biological analyses at Lyon and Paris only.

Number of Subjects: 62 patients (31 per group). Duration: Inclusion (24 months), individual participation (3 months), total study (27 months).

Locations: CH Le Vinatier (Lyon), CHU Nantes, CHU Dijon, CHU Clermont Ferrand, CH Rouen, GHU Neurosciences Paris.

Benefit-Risk Ratio: Pioneering study on tDCS in DS, aiming for a safe alternative to current treatments and a better understanding of neurobiological mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Patient with Down syndrome
* Age > 18
* Diagnosis of Major Depressive Disorder MDD with catatonic symptoms according to the DSM-5 criteria
* Informed consent signed by the patient, by the patient under curatorship, or by the legal representative in the case of a patient under guardianship.
* Person affiliated to the French social security system or equivalent

Exclusion Criteria:

* Pregnancy (checked with a pregnancy test)
* Contraindication for tDCS(i.e., cochlear implant)
* Refusal of the patients or their legal representatives
* Other persons protected under the CSP (judicial safeguard, family habilitation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-09-12 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Acute changes on depressive / catatonic symptoms between D0 and D5 measured with the Bush-Francis Catatonia Rating Scale (BFCRS) | 27 months
  The primary outcome will be the acute changes in the severity of catatonic symptoms measured by the BFCRS evaluated before treatment (D0) and after the tDCS regimen (D5). The analyses will be performed on a strict intention-to-treat sample of the evaluable patients defined in the protocol as patients with a baseline assessment and at least one post-tDCS score.

SECONDARY OUTCOMES:
Changes in clinical and cognitive will be also assessed at M1 and M3, allowing the evaluation of tDCS-induced long-term effects | 27 months
  Bush-Francis Catatonia Rating Scale (BFCRS)
Changes in clinical and cognitive will be also assessed at M1 and M3, allowing the evaluation of tDCS-induced long-term effects | 27 months
  Montgomery-Åsberg Depression Rating Scale (MADRS)
Changes in clinical and cognitive will be also assessed at M1 and M3, allowing the evaluation of tDCS-induced long-term effects | 27 months
  Unified Parkinson's Disease Rating Scale (UPDRS)
Changes in clinical and cognitive will be also assessed at M1 and M3, allowing the evaluation of tDCS-induced long-term effects | 27 months
  Severe Impairment Battery scale (SIB)

CONTACTS AND LOCATIONS:
Overall Officials: CAROLINE C DEMILY, MD PhD HDR, Principal Investigator — HOPITAL VINATIER

IPD SHARING:
Plan to Share IPD: No